CLINICAL TRIAL: NCT02125799
Title: A Pilot Trial on the Effectiveness and Tolerability of Accelerated High Frequency Repetitive Transcranial Magnetic Stimulation for Treating Resistant Major Depression
Brief Title: Accelerated rTMS for Treatment-Resistant Major Depression
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Douglas Mental Health University Institute (Other)
Responsible Party: Principal Investigator, MARCELO T. BERLIM, Director, Neuromodulation Research Clinic, Douglas Mental Health University Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ERB12/38; IRB12/38 (Other: Douglas Institute - Institutional Review Board)
Record Dates: First submitted 2014-04-25; First posted 2014-04-29 (Estimated); Last update posted 2014-10-06 (Estimated); Status verified 2014-10

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Accelerated HF-rTMS (Experimental): Twice daily rTMS sessions involving 10 Hz in 75 trains of 4 seconds duration, with 26 seconds intertrain intervals (6,000 pulses per day) at 120% of the resting motor threshold.
  Interventions: Device: Accelerated HF-rTMS (Magstim Rapid 2 stimulator)

INTERVENTIONS:
Device: Accelerated HF-rTMS (Magstim Rapid 2 stimulator) — Twice daily rTMS sessions involving 10 Hz in 75 trains of 4 seconds duration, with 26 seconds intertrain intervals (6,000 pulses per day) at 120% of the resting motor threshold.

SUMMARY:
High frequency repetitive transcranial magnetic stimulation (HF-rTMS) has shown safety and efficacy for treatment-resistant depression, but requires daily treatment for 4-6 weeks. Accelerated HF-TMS (aHF-rTMS), in which all treatments are delivered in less time, would have significant advantages in terms of access, patient acceptance and costs. In the present open label trial the investigators intend to assess the effectiveness and acceptability of a novel aHF-rTMS protocol (i.e., 2 daily sessions over 2 consecutive weeks; 6,000 pulses per day). For this, depressed outpatients will receive the aHF-rTMS protocol and will be assessed at baseline and at weeks 3 and 9 with several clinician- and patient- reported measures as well as with computerized neurocognitive tests.

ELIGIBILITY:
Inclusion Criteria:

* Presence of a current major depressive disorder (according to the DSM-IV-TR) that has not improved after ≥ 2 adequate antidepressant trial(s) in the current episode;
* Baseline score ≥ 13 on the QIDS-C
* Stable medication regimen (>= 4 weeks) prior to study enrolment

Exclusion Criteria:

* Psychotic features in the current episode
* Lifetime history of psychotic disorders and/or bipolar I or II disorders
* Substance or alcohol abuse/dependence in the past 6 months
* Lifetime history of a major neurological disease (e.g., Parkinson's, stroke)
* Uncontrolled medical disease (e.g., cardiovascular, renal)
* Pregnancy and/or lactation
* Presence of a specific contraindication for rTMS (e.g., personal history of epilepsy, metallic head implant)
* Hearing loss

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Quick Inventory of Depressive Symptomatology - Clinician Version | Week 3
  Response to treatment is defined as a ≥ 50% reduction in the scores of the QIDS-C. Remission is defined as a QIDS-C score ≤ 5.

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Berlim, MD, MSc, Principal Investigator — McGill University - Dept of Psychiatry
Locations (1):
- Douglas Mental Health University Institute, Montreal, Quebec, Canada